CLINICAL TRIAL: NCT01450267
Title: Randomized, Single Blind, Controlled Trial of Inhaled Glutathione Versus Placebo in Patients With Cystic Fibrosis
Brief Title: Inhaled Glutathione (GSH) Versus Placebo in Cystic Fibrosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Serafino A. Marsico (Other)
Collaborators: Federico II University (Other)
Responsible Party: Sponsor-Investigator, Serafino A. Marsico, Professor of Respiratory Diseases, University of Campania Luigi Vanvitelli
Organization: University of Campania Luigi Vanvitelli (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FARM7K7XZB
Record Dates: First submitted 2011-09-30; First posted 2011-10-12 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Glutathione
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiological solution (Placebo Comparator)
  Interventions: Drug: Physiological solution
- Reduced Inhaled Glutathione (Experimental)
  Interventions: Drug: Inhaled Reduced Glutathione

INTERVENTIONS:
Drug: Inhaled Reduced Glutathione — 10 mg/kg, twice daily, 12 months
  Other Names: GSH
  Arms: Reduced Inhaled Glutathione
Drug: Physiological solution — 0,13 ml/kg body weight, twice daily, 12 months
  Other Names: 0,9% sodium chloride sterile solution,
  Arms: Physiological solution

SUMMARY:
Cystic fibrosis (CF) is the most common inherited disease among the Caucasian population with considerable morbidity and reduced life expectancy.

Excessive oxidants released by activated inflammatory cells and persisting infections are considered the main mechanism of damage of respiratory epithelium in CF.Glutathione (GSH) represents the first-line defence of the lung against oxidative stress-induced cell injury; however, a depletion of its levels has been observed in the airways of patients affected by CF. In vitro studies have showed that CFTR protein plays a pivotal role in transmembrane glutathione transport. Therapeutic approaches with inhaled GSH could improve the reduced lung antioxidant capacity in order to counterbalance the oxidant stress linked to the chronic airway inflammation and bacterial infection.

Primary objective of the study is to investigate whether a 12 months treatment with inhaled GSH can improve airway obstruction in CF patients. Secondary objectives include the effects of GSH therapy on exercise capacity, body mass index (BMI), respiratory symptoms, quality of life, frequency of pulmonary exacerbations, hospital admissions, and antibiotic administration. Moreover the study will evaluate the effect of GSH therapy on markers of oxidative stress in exhaled breath condensate (EBC) and in serum, and on inflammatory markers on brushed nasal epithelial cells.

DETAILED DESCRIPTION:
150 eligible patients will be enrolled on the basis of inclusion criteria. Patients will be divided in two groups: 1) Group 1 age between 6 and 18 years; 2) Group 2 older than 18 years. Patients will be randomly assigned to the treatment or placebo arm.Patients randomized in the GSH arm will receive a dosage of 10 mg/kg bid over a 12 months period.

Clinical visits will take place at the beginning (visit 0, enrolment visit) and after one month (visit 1), three months (visit 2), six months (visit 3) nine months (visit 4), and twelve months (visit 5, end of treatments).

Follow-up clinical visits will take place one month (visit 6), three months (visit 7), six months (visit 8) after the end of treatments.

At visit 0, all eligible patients will inhale GSH (10 mg/Kg) and a dynamic spirometry will be performed before, 10 and 60 minutes after inhalation. Patients showing a decrease in FEV1 greater than 15% after GSH inhalation will be excluded from the study.

At visit 0 and at each following visits (visit 1, 2, 3, 4, 5, 6, 7 and 8) will be performed and evaluated:

* Physical examination, measurement of vital signs, body temperature,BMI,and Spirometry;
* 6 minute walking test;
* MMRC dyspnoea scale;
* Chronic cough impact questionnaire;
* Cystic Fibrosis Quality of Life Questionnaire;
* Number of pulmonary exacerbations;
* Number and duration of hospital admissions for pulmonary exacerbations;
* Number, duration and route of administration of antibiotics;
* Blood sampling for haematological and biochemical analysis;
* Brushing of nasal epithelial cell, exhaled breath condensate with evaluation of markers of oxidative stress (H2O2), and blood sample for the measurement of markers of oxidative stress in serum will be performed in a subgroup of patients at visits 0, 3, and 5.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of cystic fibrosis documented by sweat chloride test over 60 mmol/L and/or genotype analysis;
* male and female aged older than 6 years;
* stable clinical condition;
* written informed consent.

Exclusion Criteria:

* pregnancy and fertile women taking oral contraceptives;
* cigarette smoking;
* positive culture for Burkholderia Cepacia;
* history of haemoptysis or pneumothorax;
* FEV1<= 40% of the predicted value;
* hyperresponsiveness to GSH inhalation test.

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-05 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) percent | 12 months
  Increase of at least 15% of the percent of forced expiratory volume in one second (FEV1) after GSH therapy compared to placebo

SECONDARY OUTCOMES:
Small airway function | 12 months
  It will be assessed by the flow volume curve and it will bealso evaluated after 1,3,6,and 9 months from the beginning of the treatments and after 1, 3, and 6 months from the end of the treatments
Exercise Capacity | 12 months
  It will be measured by the six minutes walking test and it will be also evaluated after 1,3,6, and 9 months from the beginning of the treatments and after 1, 3, and 6 months from the end of the treatments
BMI | 12 months
  It will be also evaluated after 1,3,6, and 9 months from the beginning of the treatments and after 1, 3, and 6 months from the end of the treatments
Dyspnoea | 12 months
  It will be assessed through the Modified Medical Research Council (MMRC) dyspnoea scale and it will be also evaluated after 1,3,6, and 9 months from the beginning of the treatments and after 1, 3, and 6 months from the end of the treatments
Cough | 12 months
  It will be assessed by the Chronic Cough Impact Questionnaire (CCIQ)and it will be also evaluated after 1,3,6, and 9 months from the beginning of the treatments and after 1, 3, and 6 months from the end of the treatments
Quality of life | 12 months
  It will be assessed according to Cystic Fibrosis Quality of Life Questionnaire (CFQoL) (not for children 6-13 years old)and it will be also evaluated after 1,3,6, and 9 months from the beginning of the treatments and after 1, 3, and 6 months from the end of the treatments
Pulmonary exacerbations | 12 months
  It will be assessed evaluating the hospital admissions and antibiotic administrations. It will be also evaluated after 1,3,6, and 9 months from the beginning of the treatments and after 1, 3, and 6 months from the end of the treatments
Markers of oxidative stress (H2O2)in serum and in exhaled breath condensate (EBC) | 12 months
  It will be measured at baseline, in the middle and at the end of the study
Epithelial inflammatory markers on brushed nasal epithelial cells | 12 months
  Epithelial tyrosine phosphorylation, p38-MAPK phosphorylation, TNF alfa release will be evaluated at baseline, in the middle and at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Serafino A Marsico, PROF, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Ospedale Monaldi, Azienda Ospedaliera Universitaria Federico II, Naples, Italy

REFERENCES:
- [Background] Griese M, Ramakers J, Krasselt A, Starosta V, Van Koningsbruggen S, Fischer R, Ratjen F, Mullinger B, Huber RM, Maier K, Rietschel E, Scheuch G. Improvement of alveolar glutathione and lung function but not oxidative state in cystic fibrosis. Am J Respir Crit Care Med. 2004 Apr 1;169(7):822-8. doi: 10.1164/rccm.200308-1104OC. Epub 2004 Jan 15. PMID 14726422
- [Background] Bishop C, Hudson VM, Hilton SC, Wilde C. A pilot study of the effect of inhaled buffered reduced glutathione on the clinical status of patients with cystic fibrosis. Chest. 2005 Jan;127(1):308-17. doi: 10.1378/chest.127.1.308. PMID 15653998
- [Background] Raia V, Maiuri L, Ciacci C, Ricciardelli I, Vacca L, Auricchio S, Cimmino M, Cavaliere M, Nardone M, Cesaro A, Malcolm J, Quaratino S, Londei M. Inhibition of p38 mitogen activated protein kinase controls airway inflammation in cystic fibrosis. Thorax. 2005 Sep;60(9):773-80. doi: 10.1136/thx.2005.042564. Epub 2005 Jun 30. PMID 15994249
- [Derived] Calabrese C, Tosco A, Abete P, Carnovale V, Basile C, Magliocca A, Quattrucci S, De Sanctis S, Alatri F, Mazzarella G, De Pietro L, Turino C, Melillo E, Buonpensiero P, Di Pasqua A, Raia V. Randomized, single blind, controlled trial of inhaled glutathione vs placebo in patients with cystic fibrosis. J Cyst Fibros. 2015 Mar;14(2):203-10. doi: 10.1016/j.jcf.2014.09.014. Epub 2014 Nov 4. PMID 25458463